CLINICAL TRIAL: NCT06922110
Title: A Multicenter, Open-label, Long-term, Safety, Tolerability, and Efficacy Study of Azetukalner in Major Depressive Disorder
Brief Title: An Open-Label Study of Azetukalner in Major Depressive Disorder
Acronym: X-NOVA-OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XPF-010-D303
Record Dates: First submitted 2025-03-20; First posted 2025-04-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Antidepressant; XEN1101; Azetukalner
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azetukalner 20 mg (Experimental)
  Interventions: Drug: Azetukalner

INTERVENTIONS:
Drug: Azetukalner — Azetukalner 20 mg taken orally once a day with food (with the evening meal when possible) for 52 weeks.

SUMMARY:
X-NOVA-OLE is a multicenter, open-label study to evaluate the long-term safety, tolerability, and efficacy of azetukalner as a monotherapy in adult participants who successfully completed an antecedent Phase 3 study of azetukalner in Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Participant successfully completed the treatment period of an antecedent azetukalner Phase 3 study in MDD.
* Participant provides written informed consent to participate in the study, is able to understand the procedures and study requirements, and agrees to abide by them.
* Participant is willing to comply with the contraception requirements.
* Male participants must agree not to donate sperm until 3 months after the last dose of study drug. Female participants must agree not to donate ova until 3 months after the last dose of study drug.

Exclusion Criteria:

* Participant met any of the withdrawal criteria, or discontinued study drug early, or was terminated early from an antecedent study.
* Participant had any protocol deviations in an antecedent azetukalner study that, in the opinion of the investigator, would preclude participation in this study.
* Participant is unable to comply with study procedures or is inappropriate for the study, as judged by the investigator.
* Participant has any medical condition, personal circumstance, or ongoing AE (from an antecedent study) that, in the opinion of the investigator, exposes the participant to unacceptable risk by participating in the study or prevents adherence to the protocol.
* Female participant who is pregnant, breastfeeding, or planning to become pregnant within 3 months after the last dose of study drug.
* Participant is planning to enter a clinical study with a different investigational drug or planning to use any experimental device for treatment of any medical condition during the study or within 28 days after completion of this study.
* Participant is judged to have a significant risk for self-harm or suicidal behavior or is considered to be an imminent danger to themself or others, as determined by the C-SSRS or in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Severity and frequency of treatment-emergent adverse events, serious adverse events, adverse events of special interest, and events of clinical interest | From the start of treatment in the open-label extension study through 8 weeks after the last dose

SECONDARY OUTCOMES:
Change from baseline in the Hamilton Depression Rating Scale, 17-Item (HAMD-17) total score over time | From baseline through the active extension treatment (Week 52)
Change from baseline in the Snaith-Hamilton Pleasure Scale (SHAPS) total score over time | From baseline through the active extension treatment (Week 52)
Change in the Clinical Global Impression of Severity (CGI-S) score over time | From baseline through the active extension treatment (Week 52)
Change from baseline in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) total score, Q-LES-Q-SF medication and life satisfaction and contentment in item scores over time | From baseline through the active extension treatment (Week 52)
Change from baseline in Sheehan Disability Scale (SDS) total score and subscale scores over time | From baseline through the active extension treatment (Week 52)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Ima Clinical Research - Phoenix, Phoenix, Arizona
  - Sanro Clinical Research Group, Llc, Bryant, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Calneuro Research Group, Inc., Los Angeles, California
  - Excell Research Inc., Oceanside, California
  - Atp Clinical Research, Orange, California
  - Nrc Research Institute, Orange, California
  - Artemis Institute For Clinical Research - San Diego, San Diego, California
  - Cenexel Cnr - Sherman Oaks, Sherman Oaks, California
  - Cenexel Cns - Torrance, Torrance, California
  - Pacific Clinical Research Management, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Pharmasouth Research, Coral Gables, Florida
  - Cns Clinical Research - Coral Springs, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Neoclinical Research, Hialeah, Florida
  - Clinical Neuroscience Solutions Inc. - Jacksonville, Jacksonville, Florida
  - Accel Research Sites - St. Petersburg-Largo, Largo, Florida
  - Harmony Clinical Research Inc, North Miami Beach, Florida
  - Clinical Neuroscience Solutions Inc. - Orlando, Orlando, Florida
  - Combined Research Orlando Phase I-Iv, Orlando, Florida
  - Panhandle Research and Medical Clinic, Pensacola, Florida
  - Advanced Discovery Research, Llc, Atlanta, Georgia
  - Synexus - Atlanta, Atlanta, Georgia
  - DelRicht Research, Atlanta, Georgia
  - Cenexel Iresearch - Atlanta, Decatur, Georgia
  - Psych Atlanta, Pc, Marietta, Georgia
  - Cenexel Iresearch - Savannah, Savannah, Georgia
  - Chicago Research Center Inc., Chicago, Illinois
  - Advanced Quality Medical Research, LLC, Orland Park, Illinois
  - Adams Clinical - Boston, Boston, Massachusetts
  - Boston Clinical Trials Llc, Boston, Massachusetts
  - Elixia MA, LLC, Springfield, Massachusetts
  - Adams Clinical - Watertown, Watertown, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Ima Clinical Research - Las Vegas, Las Vegas, Nevada
  - Redbird Research, Las Vegas, Nevada
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Integrative Clinical Trials, Llc, Brooklyn, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Insight Clinical Trials Llc, Independence, Ohio
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Delricht Research - Plano, Plano, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No